CLINICAL TRIAL: NCT06186856
Title: Epidemiological Data on Mast Cell Pathologies in France
Acronym: DATAMAST
Status: Recruiting | Type: Observational
Sponsor: Imagine Institute (Other)
Responsible Party: Sponsor
Other Study IDs: HJ-22-DATAMAST
Record Dates: First submitted 2023-11-21; First posted 2024-01-02 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Mast Cell Disorder
Keywords: Mast Cell Disease; Mastocytosis; mast cell-associated diseases
MeSH Terms: conditions — Mastocytosis; Mast Cell Activation Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients

SUMMARY:
Mast cell disorders constitute a heterogeneous group of diseases, including :

* mastocytosis, i.e. cutaneous, indolent and severe forms of the disease, such as aggressive mastocytosis and mast cell leukemia) ;
* mast cell-associated diseases such as mast cell activation syndrome (idiopathic, secondary or clonal), affecting both children and adults.

No epidemiological data are currently available in France.

In France, medical care of mast cell disorders is mainly provided by a rare disease network (CEREMAST), whose CRMR is located at the Necker Enfants Malades hospital in Paris. A total of 20 centers are located throughout France.

Our aim is to use this network to study patients suffering from these diseases. The overall aim of the study is to improve the understanding, diagnosis, prognosis, recognition and management of patients with mastocytosis.

ELIGIBILITY:
Inclusion Criteria:

1. Children from birth and adults of any age
2. With one of the following mast cell diseases:

   * Mastocytoses (cutaneous, systemic and sarcomas) Defined according to the WHO 2016 classification
   * Mast cell activation syndromes (idiopathic, secondary and clonal)
   * Other mast cell activation disorders (MCAD-NOS), Defined according to the Vienna classification
   * Pre-mastocytosis or MMC (1 to 2 criteria according to WHO 2016 classification).
3. Managed in France in a rare disease reference, constitutive or competence center (CEREMAST) with DGOS labelization.

Exclusion Criteria:

1. Opposition of the patient or his/her parents to participation in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient with mast cell diseases, managed in France in a rare disease reference center CEREMAST.
  13000 pateints estimated.
Sampling Method: Non-Probability Sample
Enrollment: 13000 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2038-12-31 (Estimated); Study Completion 2038-12-31 (Estimated)

PRIMARY OUTCOMES:
Epidemiology of mast cell disorders in France assessed by statistics on the prevalence on the various types of mast cell disorders | Data 2010 - 2038
Epidemiology of mast cell disorders in France assessed by statistics on the incidence on the various types of mast cell disorders | Data 2010 - 2038

SECONDARY OUTCOMES:
Patient characteristics | Data 2010 - 2038
  age, gender, personal and family medical history
Characteristics of mast cell disease assessed by type of disease | Data 2010 - 2038
Characteristics of mast cell disease assessed by diagnostic criteria | Data 2010 - 2038
Characteristics of mast cell disease assessed by symptoms of disease | Data 2010 - 2038
Evolution of mast cell disease assessed by progression of skin lesions | Data 2010 - 2038
Evolution of mast cell disease assessed by progression to aggressive form | Data 2010 - 2038
Evolution of mast cell disease assessed by associated hemopathy | Data 2010 - 2038
Evolution of mast cell disease assessed by appearance of new symptoms | Data 2010 - 2038
Patient follow-up assessed by occurrence of other medical events in the patient | Data 2010 - 2038
Patient follow-up assessed by overall survival | Data 2010 - 2038
Types of treatment used on mastocytosis and any associated hemopathy | Data 2010 - 2038
Tolerance of treatment used on mastocytosis and any associated hemopathy | Data 2010 - 2038
Efficacy of treatment used on mastocytosis and any associated hemopathy | Data 2010 - 2038

CONTACTS AND LOCATIONS:
Locations (20):
- France (20):
  - CHU AMIENS site sud, Amiens
  - Chu Angers, Angers
  - Chu - Besancon, Besançon
  - Chu - Caen, Caen
  - Chu - Clermont Ferrand, Clermont-Ferrand
  - CHU Grenoble, Grenoble
  - Chru Lille, Lille
  - Chu - Limoges, Limoges
  - Hospices Civils de Lyon, Lyon
  - Chu - La Timone - Marseille, Marseille
  - CHU de Montpellier, Montpellier
  - CHU de NANCY, Nancy
  - Chu - Nantes, Nantes
  - Hôpital Universitaire Pitié Salpetrière, Paris
  - Hôpital Necker-Enfants malades, Paris
  - Chu - Rennes, Rennes
  - CHU Réunion sud - Saint Pierre, Saint-Pierre
  - Chru - Strasbourg, Strasbourg
  - CHU Purpan, Toulouse
  - CHU de TOURS, Tours